CLINICAL TRIAL: NCT06540222
Title: Sustained Cord Circulation at Emergency Cesarean Section - a New Concept for Resuscitating Neonates
Brief Title: Sustained Cord Circulation at Emergency Cesarean Section
Acronym: SUCCECS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUCCECS; Dnr 2024-00276-01 (Other: The Swedish Ethical Review Authority)
Record Dates: First submitted 2024-07-03; First posted 2024-08-06 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Asphyxia Neonatorum; Fetal Hypoxia
Keywords: Emergency cesarean section; Management umbilical cord; intact cord resuscitation
MeSH Terms: conditions — Asphyxia Neonatorum; Fetal Hypoxia | interventions — Resuscitation; Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Multicenter, stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intact cord (Experimental): The neonate will be kept close to the mother with the cord intact. When in need of ventilatory support, the neonatal team will give ventilatory support with an unclamped umbilical cord, following neonatal cardiopulmonary resuscitation guidelines. Cord clamping will be performed after respiration has been established and at the earliest after three minutes and not later than five minutes.
  Interventions: Procedure: Sustained cord (≥ 180 seconds) resuscitation
- Standard care (Active Comparator): Management according to standard care, including immediate cord clamping for neonates requiring ventilatory support. In cases where ventilatory support is not necessary, cord clamping will be performed within 60 seconds of birth, adhering to established clinical guidelines for neonatal management.
  Interventions: Procedure: Routine (< 60 seconds) cord clamping

INTERVENTIONS:
Procedure: Sustained cord (≥ 180 seconds) resuscitation — Resuscitation performed in near proximity to the mother with umbilical cord uncut
  Other Names: Intact cord resuscitation; Delayed cord clamping
  Arms: Intact cord
Procedure: Routine (< 60 seconds) cord clamping — Resuscitation performed at a designated area after umbilical cord is cut
  Other Names: Immediate clamping
  Arms: Standard care

SUMMARY:
The goal of this clinical trial is to evaluate if sustained cord circulation during resuscitation improves outcomes for term neonates born by emergency Cesarean section. The main question it aims to answer is: Does sustained cord circulation reduce admission rates to neonatal care?

Researchers will compare resuscitation with an uncut umblical cord to standard resuscitation practices to see if it provides better outcomes.

Participants (term neonates born by emergency Cesarean section) will:

Receive resuscitation with either sustained cord circulation or standard care Be monitored for admission to neonatal care and other predefined health outcomes

DETAILED DESCRIPTION:
Study Title

Sustained Cord Circulation During Resuscitation of Non-Breathing Neonates Born by Cesarean Section: A Multicenter Randomized Controlled Trial

Primary Objectives:

To compare neonatal outcomes between two different approaches to resuscitation of term neonates born by CS; Intact cord resuscitation versus standard care with immediate cord clamping, and evaluate:

A composite outcome of admission to neonatal care for predefined criteria or death before admission. Predefined criteria include asphyxia at birth, respiratory distress, hypoxic ischemic encephalopathy (HIE) and hypoglycemia. Assessed within one week after birth.

Secondary Objectives: Secondary outcomes will include short and long-term neonatal outcomes, adverse maternal and neonatal outcomes, and caregivers' and staff's experiences.

Study Design: A multicenter, stepped-wedge cluster randomized trial.

Study Population: Singleton neonate born alive, gestational age ≥37 weeks, born by emergency cesarean section, epidural/spinal anesthesia. Pediatric team summoned before birth due to health concerns regarding the neonate.

Intervention: Resuscitation with intact cord circulation during 3-5 minutes. When in need of respiratory support, the neonate will be kept close to the mother with the cord intact and the placenta attached to the uterine wall. The pediatric team will give respiratory support with sustained cord circulation, following Swedish neonatal CPR guidelines. Cord clamping will be performed after respiration has been established and at the earliest after three minutes. Cord clamping will be performed at the latest at 5 minutes.

Control: Resuscitation will be performed after the cord was cut. When in need of respiratory support, the cord will be clamped immediately, and the neonate will be taken to an adjacent place for resuscitation according to Swedish neonatal CPR guidelines. Well neonates will have their cord clamped after 1 minute in accordance with national recommendations.

Power analysis: At a significant level of 0.05, the power to detect the anticipated risk reduction (15%) would be 0.88 (two-sided).

Study Duration 2025-2028

ELIGIBILITY:
Inclusion Criteria:

* Singleton neonate
* Born alive
* Gestational age ≥37 weeks
* Born by emergency cesarean section, epidural/spinal anesthesia, where the pediatric/neonatal team has been called for to attend.

Exclusion Criteria:

* Major congenital malformation that may affect resuscitation or outcome measures.
* Major genetic disorder that may affect resuscitation or outcome measures.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2200 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Composite outcome of admission to neonatal care for predefined criteria and death before admission. | At one hour after birth
  Admission to neonatal care is collected from the Swedish Neonatal Quality registry (SNQ), as are criteria for admission:• Asphyxia at birth (One-, Five- and/or Ten-minute Apgar score <4), diagnosis P21.0, P21.1A, P21.1B or P21.9.• Respiratory distress (Noted in SNQ as NAS, neonatal respiratory distress P22.8, PAS, pulmonary adaption disturbance P 22.1, RDS, respiratory distress syndrome P22.0, MAS meconium aspiration syndrome P24.0, PPHN, Persistant Pulmonary Hypertension P29.3B, or PTX, Pneumothorax P25.1).• Hypoxic-ischemic encephalopathy grade I-III, P91.6A, B, C, or X.• Hypoglycemia, P 70.4A, or B. Death of the neonate before admission is collected from Swedish pregnancy registry.
  Units of measure is dichotomous, as appearance of the diagnoses or not.

SECONDARY OUTCOMES:
Apgar score at 5 min | 5 minutes
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes, each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Less than 4 is a measure for severe asphyxia, less than 7 measure of mild asphyxia.
Apgar score at 10 min | 10 minutes
  Assessed by staff, composite of heart rate, breathing effort, skin color, muscle tone and reflexes, each sub scale 0 (absent), 1, 2 (normal). Minimum 0, maximum 10. Less than 4 is a measure for severe asphyxia, less than 7 measure of mild asphyxia.
Respiratory distress as a diagnosis after birth | One week after birth
  Having the at least one of the following diagnosis in the Swedish neonatal quality registry: NAS, neonatal respiratory distress P22.8, PAS, pulmonary adaption disturbance P 22.1, RDS, respiratory distress syndrome P22.0, MAS meconium aspiration syndrome P24.0, PPHN, Persistent Pulmonary Hypertension P29.3B, or PTX, Pneumothorax P25.1.
Hypoxic-ischemic encephalopathy as a diagnosis after birth | One week after birth
  Having the at least one of the following diagnosis in the Swedish neonatal quality registry: Hypoxic-ischemic encephalopathy grade I-III, P91.6A, B, C, or X.
Hypoglycemia as a diagnosis after birth | One week after birth
  Having the at least one of the following diagnosis in the Swedish neonatal quality registry: Hypoglycemia, P 70.4A, or B.
Duration of neonatal care | One month
  Duration of neonatal care as noted in the Swedish pregnancy register and Swedish neonatal quality registry: Aggregated as day (continuous) and ≥ 2 days, dichotomous
Death after birth but before admission to neonatal unit | One hour after birth
  Noted as dead after birth in the Swedish pregnancy register

OTHER OUTCOMES:
Neonatal outcomes - breathing | Birth to one hour
  After birth (data registered on the resuscitation chart or imported from monitor equipment):
  Initiation and establishment of breathing (Minutes and seconds)
Neonatal outcomes - temperature | Birth to six hours
  After birth (data registered on the resuscitation chart, source data sheet or imported from monitor equipment):
  Temperature (degrees Celsius)
Neonatal outcomes - interventions | Birth to one hour
  After birth (data registered on the resuscitation chart or imported from monitor equipment):
  Rate of Interventions (e.g. ventilation, intubation, chest compressions) noted on the resuscitation chart
Neonatal outcomes - heart rate | Birth to 24 hours
  After birth (data registered on the resuscitation chart or imported from monitor equipment):
  Data from Heart rate and Oxygen saturation monitoring
  Unit of measure: Heart rate
Neonatal outcomes - oxygen saturation | Birth to 24 hours
  After birth (data registered on the resuscitation chart or imported from monitor equipment):
  Data from Heart rate and Oxygen saturation monitoring
  Unit of measure: Oxygen saturation
Neonatal outcome - hyperbilirubinemia and jaundice | Birth to seven days
  Neonatal jaundice requiring phototherapy, (diagnoses reported in SPR and/or SNQ). P58.3, P59.8 (immunizations and hemolytic disorders will be excluded in this analysis)
Neonatal morbidity | Birth to one month
  During neonatal care (diagnosis from registries):
  Neonatal seizures Neonatal infection Neonatal jaundice Intracranial hemorrhage
  Unit of measure: Diagnosis occurring in Swedish Neonatal Quality registry
Maternal outcomes - maternal death | Child's birth until 6 weeks
  Maternal death, collected from SPR (O 95, O95.9, O97)
Maternal outcomes - maternal blood loss | Birth to one month
  Maternal blood loss (Amount of postpartum bleeding, ml) Severe post-partum hemorrhage (> 1000 ml and > 2000 ml)
Maternal outcomes - post-surgery infection | Birth to one month
  Maternal post-surgery infection
  Unit of measure: Diagnosis occurring in Swedish Pregnancy registry
Development assessed by ASQ at 12 months of age | 12 months
  Assessed by Ages and Stages Questionnaire (ASQ). Minimum 0, maximum 300. Consist of 30 questions answered Yes (10), Sometimes (5), Not Yet (0). Five sub scales with six questions each: Communication, Fine motor, Gross motor, Problem solving and Personal-Social. Worse outcome is considered mean minus 2 standard deviations. 'At risk' outcome is considered mean minus 1 standard deviations.
Development | 24 months
  Assessed by Ages and Stages Questionnaire (ASQ). Minimum 0, maximum 300. Consist of 30 questions answered Yes (10), Sometimes (5), Not Yet (0). Five sub scales with six questions each: Communication, Fine motor, Gross motor, Problem solving and Personal-Social. Worse outcome is considered mean minus 2 standard deviations. 'At risk' outcome is considered mean minus 1 standard deviations.
Development | 36 months
  Assessed by Ages and Stages Questionnaire (ASQ). Minimum 0, maximum 300. Consist of 30 questions answered Yes (10), Sometimes (5), Not Yet (0). Five sub scales with six questions each: Communication, Fine motor, Gross motor, Problem solving and Personal-Social. Worse outcome is considered mean minus 2 standard deviations. 'At risk' outcome is considered mean minus 1 standard deviations.
Development | 48 months
  Assessed by Ages and Stages Questionnaire (ASQ). Minimum 0, maximum 300. Consist of 30 questions answered Yes (10), Sometimes (5), Not Yet (0). Five sub scales with six questions each: Communication, Fine motor, Gross motor, Problem solving and Personal-Social. Worse outcome is considered mean minus 2 standard deviations. 'At risk' outcome is considered mean minus 1 standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Andersson, MD PhD, Principal Investigator — Region Skåne, Lund University; Jenny Svedenkrans, MD PhD, Principal Investigator — Karolinska University Hospital, Karolinska Institutet
Locations (12):
- Sweden (12):
  - Östra sjukhuset - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Hallands sjukhus, Halmstad, Halmstad
  - Universitetssjukhuset i Linköping, Linköping
  - Skånes Universitetssjukhus, Lund
  - Skånes Universitetssjukhus, Malmö, Malmo
  - Universitetssjukhuset Örebro, Örebro
  - BB Stockholm, Stockholm
  - Danderyds sjukhus, Stockholm
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
  - Karolinska Universitetssjukhuset, Solna, Stockholm
  - Södersjukhuset - Sachsska barn- och ungdomssjukhuset, Stockholm
  - Norrlands universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: No
At present we are not allowed to share anonymized data extracted from Swedish medical health registers.

REFERENCES:
- [Background] Ekelof K, Saether E, Andersson O, Svedenkrans J, Linden K. pre-SUCCECS: Lessons learned from implementing resuscitation and stabilisation with an intact cord during caesarean sections - Focus group discussions with implementation teams. Sex Reprod Healthc. 2025 Sep;45:101114. doi: 10.1016/j.srhc.2025.101114. Epub 2025 May 26. PMID 40479951
- [Background] Alikhani VS, Thies-Lagergren L, Svedenkrans J, Elfvin A, Bolk J, Andersson O. Stabilisation and resuscitation with intact cord circulation is feasible using a wide variety of approaches; a scoping review. Acta Paediatr. 2023 Dec;112(12):2468-2477. doi: 10.1111/apa.16985. Epub 2023 Sep 28. PMID 37767916
- See also: Homepage of the SUCCECS study (in Swedish) — https://www.succecs.se/